CLINICAL TRIAL: NCT00550368
Title: Effect of Gastric Acid and H. Pylori Infection on Infection With Enteropathogenic E. Coli
Brief Title: Clinical Experiment of Helicobacter Pylori Transmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Julie Parsonnet, Principle Investigator, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 688; NCT00549224 (obsolete NCT alias)
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-10

CONDITIONS: Infection; Achlorhydria
MeSH Terms: conditions — Infections; Achlorhydria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Helicobacter pylori negative (Experimental): Persons who tested negative for H. pylori by both serology and Urea breath test. All participants will receive the Biological intervention: Enteropathogenic E. coli.
  Interventions: Biological: Biological intervention: Enteropathogenic E. coli
- Helicobacter pylori positive (Experimental): Persons who tested positive for H. pylori by both serology and Urea breath test. All participants will receive the Biological intervention: Enteropathogenic E. coli.
  Interventions: Biological: Biological intervention: Enteropathogenic E. coli

INTERVENTIONS:
Biological: Biological intervention: Enteropathogenic E. coli — 5x10^8 or 1x10^9 organisms of EPEC were administered to all participants.

SUMMARY:
The study proposes to test whether chronic infection with Helicobacter pylori protects individuals from symptomatic infection with enteropathogenic E. coli. The study will also evaluate the effect of gastric acidity in this relationship.

DETAILED DESCRIPTION:
Because H. pylori is an enteric infection, its prevalence may be linked to exposure to other enteric pathogens. Results of observational studies on the association between H. pylori and gastroenteritis, however, have been conflicting. Some have shown increased incidence of diarrhea in children with H. pylori infection, with one study attributing 11% of diarrhea cases to H. pylori. Other studies found no association, and still others found a protective effect of H. pylori against gastroenteritis. Dissecting out confounding from true physiological associations can be difficult in observational studies. To better elucidate the association between H. pylori and gastroenteritis, we performed a direct challenge experiment with a well-characterized gastrointestinal pathogen, enteropathogenic Escherichia coli (EPEC). EPEC is a leading cause of infantile gastroenteritis in the world and has a long history of safe use in human experiments. It is also acid sensitive: in our laboratory less than 0.001% of inoculated EPEC organisms survived at pH 2.5. Our goal was to test the hypothesis that chronic infection with H. pylori increases the risk of diarrheal illness after direct challenge with EPEC.

ELIGIBILITY:
Inclusion Criteria:Healthy Exclusion Criteria:prior gastrointestinal disease prior treatment of H. pylori infection immune suppression or deficiency history of cancer, diabetes, or other co-morbidity

Ages: 35 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2005-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Parsonnet, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited for the study from 2005 to 2008. Enrollment began 6/2005 and ended 5/2008. Healthy individuals were sought with no chronic medical conditions or symptoms.
Pre-assignment Details: Participants were assigned to one of two groups: Helicobacter pylori positive, or Helicobacter pylori negative. Assignment was based on results of H. pylori serology and Urea Breath Test. Test results had to be concordant for group assignment.
Groups:
- H. Pylori Negative: Participants who tested negative for H. pylori infection.
- H. Pylori Positive: Participants who tested H. pylori positive
Period: Overall Study
Arm/Group | H. Pylori Negative | H. Pylori Positive
Started | 26 | 19
Completed | 26 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H. Pylori Negative | H. Pylori Positive | Total
Number analyzed (Participants) | 26 | 19 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (7.3) | 49.4 (6.7) | 48.6 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 12 | 17
  Not Hispanic or Latino | 21 | 7 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 21 | 13 | 34
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 27 (4.5) | 28.7 (3.8) | 27.7 (4.3)
Gastric pH, Median [Median (Full Range); unit: units on a scale] | 1.5 [1.1 to 6.8] | 1.6 [1.2 to 7.5] | 1.5 [1.1 to 7.5]
Hypochlorhydric [Number; unit: participants] | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Development of Diarrhea
Time Frame: 48 hours
Measure: Number; unit: participants
Arm/Group | H. Pylori Negative | H. Pylori Positive
Number analyzed (Participants) | 26 | 19
participants | 5 | 6

2. Secondary Outcome: Intensity of Gastrointestinal Symptoms
Description: Composite gastrointestinal symptom score was on a scale from 0 (no symptoms) to 15 (severe symptoms). This composite was the sum of 5 self-reported, symptom scores, each ranging from 0 (none) to 3 (severe). The self-reported symptoms that subjects scored were: malaise, headache, nausea, vomiting, and loose stool.
Time Frame: 48 hours
Measure: Median (Full Range); unit: units on a scale
Arm/Group | H. Pylori Negative | H. Pylori Positive
Number analyzed (Participants) | 26 | 19
units on a scale | 3 [0 to 15] | 3 [0 to 15]

ADVERSE EVENTS:
Time Frame: Participants were monitored for 48 hours as inpatients following ingestion of 5x10^8 or 1 x10^9 organisms of Enteropathogenic E. coli. After discharge, participants were further followed for 4 weeks from the time of discharge from the hospital.
Arm/Group | H. Pylori Negative | H. Pylori Positive
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/19
Other Adverse Events (participants affected / at risk) | 0/26 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No